CLINICAL TRIAL: NCT01111708
Title: Clinical Outcome After Close Rectal Ileo Pouch Anal Anastomosis for Colitis Ulcerosa Compared to the Ileo Neo Rectal Anastomosis and the Ileo Pouch Anal Anastomosis
Brief Title: Clinical Outcome After Close Rectal Ileo Pouch Anal Anastomosis for Colitis Ulcerosa(CU)
Acronym: CR-IPAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Nijmegen (Other)
Responsible Party: Sharonne de Zeeuw, Academic University of Nijmegen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Close Rectal - IPAA
Record Dates: First submitted 2010-04-26; First posted 2010-04-27 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Close Rectal-Ileo Pouch Anal Anastomosis (Experimental)
  Interventions: Procedure: Close Rectal Dissection - IPAA
- Conventional Ileo Pouch Anal Anastomosis (Active Comparator)
  Interventions: Procedure: Close Rectal Dissection - IPAA
- Ileo Neo Rectal Anastomosis (Active Comparator)
  Interventions: Procedure: Close Rectal Dissection - IPAA

INTERVENTIONS:
Procedure: Close Rectal Dissection - IPAA — Comparison between conventional IPAA and Close Rectal IPAA and INRA after (sub)total proctocolectomy for Ulcerative colitis
  Other Names: INRA, IPAA, restorative surgery

SUMMARY:
The purpose of this study is to investigate a new technique: Close Rectal Dissection (CRD) as restorative surgery for Ulcerative Colitis patients: the Close Rectal Ileo Pouch Anal Anastomosis (CR-IPAA). Clinical outcome and quality of life will be compared to the conventional Ileo Pouch Anal Anastomosis (C-IPAA) and the Ileo Neo Rectal Anastomosis (INRA).

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is characterized by recurring episodes of inflammation limited to the mucosal layer of the colon. The surgery rate after 10 years is 30%. After (sub)total colectomy with end ileostoma patients have a choice for restorative surgery. The conventional ileo pouch anal anastomosis (C-IPAA) is the gold standard of reconstructive surgery. This is al well established technique, but still carries a significant morbidity-rate. The recent studied ileo neo rectal anastomosis (INRA) has shown to reduce reservoir-related complications with a similar functional outcome, but is a very laborious technique. Therefore, we want to investigate an alternative technique: the Close Rectal Ileo Pouch Anal Anastomosis (CR-IPAA). The CR-IPAA is conducted in the nonanatomic perimuscular plane, resulting in a reduction of reservoir-related complications. After the close rectal dissection an ileo-anal pouch anastomosis will be constructed in a similar way. The close rectal dissection (CRD) is very laborious and has therefore never been developed extensively. But recent technical development of electrothermal bipolar vessel sealer (EBVS ) and ultrasound dissection have enhanced the CRD technique enormously. This brought along new interest in the CRD and justifies the research of its application.

ELIGIBILITY:
Inclusion Criteria:

* UC patients with the CRD procedure with written informed consent.
* Age, sex and disease specific matched control group op UC-IPAA patients with written informed consent.

Exclusion Criteria:

* Pregnancy
* Malignancy
* Psychiatric disease or inability to assess follow-up

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
To determine the clinical outcome (functional outcome and morbidity) after CR-IPAA compared to C-IPAA and INRA and to compare quality of life in these three different groups. | 1 year

SECONDARY OUTCOMES:
Secondary objectives are the inflammatory responses (pouchitis), ano-rectal function, meso-rectal development on MRI, endoscopy results and histopathology. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kees v Laarhoven, prof. dr., Study Director — Radboud University Medical Center
Locations (1):
- Universitair Medical Centre St. Radboud, Nijmegen, Gelderland, Netherlands